CLINICAL TRIAL: NCT06647056
Title: Evaluation of the Effect of a Single Dose of Psilocybin on Neural Correlates of Cognitive Control in Patients With Psychogenic Nonepileptic Seizures
Acronym: CRIPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2022-2/IC01
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Psychogenic Nonepileptic Seizures; Psilocybin
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with PNES (Experimental)
  Interventions: Drug: Psilocybin; Other: MRI

INTERVENTIONS:
Drug: Psilocybin — Administration of psilocybin 25 mg
Other: MRI — Two standard MRI + fMRI scans before (D-3) and after (D5) treatment

SUMMARY:
Psychogenic non-epileptic seizures (PNES) are functional paroxysmal motor disorders that may be clinically suggestive of epilepsy but are not associated with the electroencephysiological and electroencephalographic changes of epilepsy. Thus, hyper-connectivity of the regions of the default mode network (DMN) linked to executive control could be involved in the impairment of cognitive control capacities in patients suffering from PNES. Also, the HYCORE study (NCT02329626), showed that dysregulation of frontal regions involved in attentional and emotional regulation is correlated with motor symptoms in patients with functional neurological disorders.

The researchers of this study hypothesized that psilocybin would improve cognitive control in patients with PNES.

ELIGIBILITY:
Inclusion Criteria:

* Euthymic patient according to the MINI questionnaire.
* Diagnosis of PNES confirmed by video-EEG, progressing for more than 3 months, and meeting DSM5 criteria.
* Normal brain MRI during the assessment as part of routine care
* No contraindication to stopping any antidepressant treatment for a fortnight (or 5 weeks for fluoxetine) prior to the administration of psilocybin. Other psychotropic treatments will not be interrupted.
* Patient must have given their free and informed consent and signed the consent form
* Patient must be a member of beneficiary of a health insurance plan
* Patient available for a total of 6 months follow-up.
* Good physical health and absence of unstable medical pathology. These pathologies include cardiovascular co-morbidities: history of stroke, myocardial infarction, heart failure, arrhythmia, uncontrolled hypertension (greater than 165/95 mmHg at screening); organic epileptic syndrome and active neurological comorbidities; endocrine pathologies (dysthyroid and adrenal insufficiency, type 1 diabetes or insulin-requiring type II diabetes, history of severe hypoglycaemia requiring hospital treatment); considerable impairment of liver function; glaucoma; symptomatic prostatic hypertrophy or bladder neck obstruction.
* Ability to understand and speak French

Exclusion Criteria:

* Serious risk of suicide according to the clinician opinion.
* High risk of adverse emotional or behavioural reaction as clinically assessed by the investigator (e.g. severe personality disorder, antisocial behaviour, severe current stress factors, lack of consequent social support).
* Active dependence on a substance according to the MINI questionnaire (excluding tobacco).
* Psychotropic treatment (anxiolytics, antipsychotics, hypnotics) modified in the last month.
* Patient with intellectual disability.
* A lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder or psychosis not otherwise specified.
* Family history of schizophrenia, schizoaffective disorder or type 1 bipolar disorder in first or second degree relatives.
* Any unstable disease or physical condition determined by history or laboratory tests (ECG, blood tests at inclusion). These conditions include cardiovascular co-morbidities: history of stroke, myocardial infarction, heart failure, arrythmia, uncontrolled hypertension (greater than 165/95 mmHg at screening); organic epileptic syndrome and active neurological comorbidities; endocrine pathologies (dysthyroid and adrenal disorders, type I diabetes or insulin-requiring type II diabetes, history of severe hypoglycaemia requiring hospital treatment); considerable impairment of liver function; glaucoma, symptomatic prostatic hypertrophy or bladder neck obstruction.
* Presence of neurological comorbidities.
* Medical conditions that would preclude safe participation in the trial; for example: considerable impairment of liver function, coronary artery disease, history of arrythmia, heart failure, uncontrolled hypertension (greater than 165/95 mmHg at screening). History of stroke, severe asthma, hyperthyroid, narrow angle glaucoma, uncontrolled type I or type II diabetes or history of ketoacidosis, hyperglycaemic coma or severe hypoglycaemia with loss of consciousness.
* Participants planning to donate sperm within three months of psilocybin administration.
* Participants having sexual intercourse that could lead to pregnancy and who do not agree to use a highly effective contraceptive method (contraceptive ring, surgical contraception, implant, patch, contraceptive pill, male and female condoms, IUD) throughout their participation in the study and for at least three months after administration of psilocybin.
* Positive serum pregnancy test at inclusion for participants of childbearing age NB: serum pregnancy test will be performed prior to administration of psilocybin.
* Contraindications to magnetic resonance imaging.
* Allergy, hypersensitivity or other adverse reaction to previous use of psilocybin or other hallucinogens.
* Consumption of hallucinogenic substances (excluding cannabis) more than 10 times in a lifetime or in the last 2 months, regardless of frequency.
* Use of medication likely to interfere with the effects of psychedelics.
* Regular consumption of alcoholic beverages (>20 drinks/week).
* Any other major clinically considerable concomitant disease which, in the opinion of the investigator, may interfere with the interpretation of the results of the study or constitute a risk to the health of the participant, should they take part in the study.
* Patient with a prolonged QTc interval (interval >450 ms for men and >470 ms for women)
* Patient taking part in an interventional drug study.
* Patient in a period of exclusion determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Patient to whom it is impossible to communicate informed information
* Patient with a positive pregnancy test prior to psilocybin administration.
* Any patient who has been hospitalised on an outpatient or inpatient basis between the date of inclusion and the administration of psilocybin.
* Any patient who has made a known, interrupted or aborted suicide attempt between the date of inclusion and the administration of psilocybin.
* Any patient who has expressed suicidal ideation associated with the planning of a suicidal act (active suicidal ideation) between the date of inclusion and the administration of psilocybin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Emotional distraction in PNES patients receiving psilocybin | Three days before psilocybin treatment
  Fluctuation du signal BOLD (Blood-oxygen level dependence) during a Go-No Go test
Emotional distraction in PNES patients receiving psilocybin | Five days after psilocybin treatment
  Fluctuation du signal BOLD (Blood-oxygen level dependence) during a Go-No Go test

SECONDARY OUTCOMES:
Resting-state activity in brain regions involved in cognitive control in PNES patients receiving psilocybin | Three days before psilocybin treatment
  Fluctuation of the BOLD (Blood-oxygen level dependent) signal for each independent component (Image grey levels).
Resting-state activity in brain regions involved in cognitive control in PNES patients receiving psilocybin | Five days after psilocybin treatment
  Fluctuation of the BOLD (Blood-oxygen level dependent) signal for each independent component (Image grey levels).
Resting-state activity in brain regions of the default mode network (DMN) in patients with PNES receiving psilocybin. | Three days before psilocybin treatment
  Blood-oxygen level dependent (BOLD) signal synchronisation levels in brain regions DMN (grey levels of the image).
Resting-state activity in brain regions of the default mode network (DMN) in patients with PNES receiving psilocybin. | Five days after psilocybin treatment
  Blood-oxygen level dependent (BOLD) signal synchronisation levels in brain regions DMN (grey levels of the image).
Cognitive control abilities in patients with PNES receiving psilocybin | Three days before psilocybin treatment
  emotional Go-No Go error rate (%)
Cognitive control abilities in patients with PNES receiving psilocybin | Five days after psilocybin treatment
  emotional Go-No Go error rate (%)
Cognitive control abilities in patients with PNES receiving psilocybin | Three days before psilocybin treatment
  neutral Go-No Go task response latency (ms)
Cognitive control abilities in patients with PNES receiving psilocybin | Five days after psilocybin treatment
  neutral Go-No Go task response latency (ms)
Number of PNES over a 3-month period in patients with PNES receiving psilocybin | Day 0
  Number
Number of PNES over a 3-month period in patients with PNES receiving psilocybin | Month 3
  Number
Functional impact of PNES in patients with PNES receiving psilocybin | Three days before psilocybin treatment
  Clinical Global Impression: Score 0-7; cut-off: 4 = unchanged or worse and the secondary effects take over the therapeutic effects
Functional impact of PNES in patients with PNES receiving psilocybin | Five days after psilocybin treatment
  Clinical Global Impression: Score 0-7; cut-off: 4 = unchanged or worse and the secondary effects take over the therapeutic effects
Functional impact of PNES in patients with PNES receiving psilocybin | Month 1
  Clinical Global Impression: Score 0-7; cut-off: 4 = unchanged or worse and the secondary effects take over the therapeutic effects
Functional impact of PNES in patients with PNES receiving psilocybin | Month 3
  Clinical Global Impression: Score 0-7; cut-off: 4 = unchanged or worse and the secondary effects take over the therapeutic effects
Dissociative symptoms in patients with PNES receiving psilocybin | Three days before psilocybin treatment
  Dissociation Experience Scale: Score 0-100; cut-off: 30 or more shows the presence of dissociative troubles.
Dissociative symptoms in patients with PNES receiving psilocybin | Five days after psilocybin treatment
  Dissociation Experience Scale: Score 0-100; cut-off: 30 or more shows the presence of dissociative troubles.
Dissociative symptoms in patients with PNES receiving psilocybin | Month 1
  Dissociation Experience Scale: Score 0-100; cut-off: 30 or more shows the presence of dissociative troubles.
Dissociative symptoms in patients with PNES receiving psilocybin | Month 3
  Dissociation Experience Scale: Score 0-100; cut-off: 30 or more shows the presence of dissociative troubles.
Tolerance of psilocybin in patients with PNES receiving psilocybin | Day 0
  5-Dimensional Altered States of Consciousness Rating Scale: Score 0-100; more than 25 = higher probability to have a dissociative trouble.
Tolerance of psilocybin in patients with PNES receiving psilocybin | Five days after psilocybin treatment
  5-Dimensional Altered States of Consciousness Rating Scale: Score 0-100; more than 25 = higher probability to have a dissociative trouble.
Tolerance of psilocybin in patients with PNES receiving psilocybin | Month 1
  5-Dimensional Altered States of Consciousness Rating Scale: Score 0-100; more than 25 = higher probability to have a dissociative trouble.
Tolerance of psilocybin in patients with PNES receiving psilocybin | Month 3
  5-Dimensional Altered States of Consciousness Rating Scale: Score 0-100; more than 25 = higher probability to have a dissociative trouble.

CONTACTS AND LOCATIONS:
Overall Officials: Ismaël CONEJERO, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No